CLINICAL TRIAL: NCT04459819
Title: Monocentric, Observational, Retrospective Study on Respiratory Physiotherapy in Severe COVID-19 Patients: the FTR-COVID Study.
Brief Title: Respiratory Physiotherapy in Severe COVID-19 Patients
Acronym: FTR-COVID
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: FTR-COVID
Record Dates: First submitted 2020-06-27; First posted 2020-07-07 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: ICU; Respiratory Physiotherapy; Early Rehabilitation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Respiratory physiotherapy — Respiratory physiotherapy consists of:
  * early mobilization (passive and active mobilization, muscle-strengthening exercises, mobilization out of bed, standing, walking, ADL)
  * patients positioning
  * non-invasive mechanical ventilation / CPAP
  * tracheostomy management
  * invasive mechanical ventilation weaning
  * airway clearance
  * oxygen titration

SUMMARY:
COVID-19 is an infectious disease caused by SARS-CoV2 virus. COVID-19 patients can develop a severe disease that can lead to hypoxic respiratory failure and acute respiratory distress syndrome (ARDS). Severe patients can require access to intensive care unit (ICU). Early rehabilitation is known to be effective in critically ill patients and in ARDS.

The role of respiratory physiotherapy in critical COVID-19 patients is still unclear.

The aim of this study is to describe the bundle and the timing of respiratory physiotherapy used with severe COVID-19 patients from ICU to hospital discharge. Functional condition of patients at discharge will be assessed and described.

DETAILED DESCRIPTION:
COVID-19 is an infectious disease caused by SARS-CoV2 virus, that first appeared in China in 2019 and in Italy in February 2020.

Approximately 80% of people infected with COVID-19 have mild to moderate disease with few symptoms, while more than 10% develop a severe disease that can lead to hypoxic respiratory failure and acute respiratory distress syndrome (ARDS). Severe patients can require access to intensive care unit (ICU) needing invasive mechanical ventilation (IMV) and hospitalization for a long period.

Early rehabilitation is known to be effective in critically ill patients and in ARDS, to reduce functional impairment due to the prolonged stay in ICU. Many works demonstrated that early rehabilitation programs in ICU correlated with faster recovery and discharge at home of ARDS patients and better outcomes in the walking test at discharge from the hospital.

Due to the recent development of COVID-19, few data and guidelines to menage severe COVID-19 patients are available and the role of respiratory physiotherapy is still unclear.

The aim of this study is to describe the bundle and the timing of respiratory physiotherapy used with severe COVID-19 patients from ICU to hospital discharge. Functional condition of patients at discharge will be assessed and described.

ELIGIBILITY:
Inclusion Criteria:

* Having laboratory confirmed COVID-19 pneumonia
* Developed hypoxemic acute respiratory failure (hARF) requiring access to ICU
* Treated by respiratory physiotherapists during the hospitalization period

Exclusion Criteria:

* Previously documented neurological or neuromuscular diseases
* Passed over 1 month in bed before COVID-19 diagnosis
* Documented cognitive impairment (mini mental state examination <24)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will study patients accessing acute hospital ICU with hypoxemic acute respiratory failure (hARF) due to laboratory confirmed COVID-19 pneumonia form March 1st to May 1st, that were treated by respiratory physiotherapists during the whole hospitalization period.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Number of physiotherapy treatments | Through study completion, an average of 60 days
  Total number of physiotherapy treatments performed on patients during hospitalization
Type of physiotherapy treatments | Through study completion, an average of 60 days
  Number of each activity performed on patients among early mobilization, positioning, Uso of non invasive ventilation (NIV) and/or continuous positive airway pressure (CPAP), oxygen titration, airway clearance.
Time of the first physiotherapy treatment | From patient intubation to first time patient was treated by a physiotherapist; up to 60 days
  Median number of days from patients intubation to the first physiotherapy treatment

SECONDARY OUTCOMES:
First time standing | From patient intubation to first time standing; up to 60 days
  Median number of days from patients intubation to standing
First time walking | From patient intubation to first time walking; up to 60 days
  Median number of days from patients intubation to walking
First time sitting out of bed | From patient intubation to first time sitting out of bed; up to 60 days
  Median number of days from patients intubation to sitting out of bed
6 minutes walking test (6MWT) | Assessed when patients are discharged from the hospital; up to 60 days
  Median distance (metres) obtained at the 6MWT
1 minute sit-to-stand test (1m-STST) | Assessed when patients are discharged from the hospital; up to 60 days
  Median number of sit-to-stand repetitions obtained
Upper extremity muscles strength | Assessed at 2 time points, when patients are discharged from ICU and when patients are discharged from the hospital; up to 60 days.
  Median upper extremity muscle strength measured by the Medical Research Council sum score (MRC-SS). The muscle scale grades muscle power on a scale of 0 (no visible muscle contraction) to 5 (active movement against full resistance). The movement tested are wrist flexion, forearm flexion and shoulder abduction.
Lower extremity muscles strength | Assessed at 2 time points, when patients are discharged from ICU and when patients are discharged from the hospital; up to 60 days.
  Median lower extremity muscle strength measured by the Medical Research Council sum score (MRC-SS). The muscle scale grades muscle power on a scale of 0 (no visible muscle contraction) to 5 (active movement against full resistance). The movement tested are ankle dorsiflexion, knee extension and hip flexion.
Functional independence in ADL | Assessed when the patient is discharged from the hospital; up to 60 days.
  Median score obtained th the Barthel Index for Activities of Daily Living (ADL). The Barthel Index measures functional independence in ADL. Scores range from 0 to 100, with higher scores indicating greater independence in ADL.
ICU stay length | From ICU admission to ICU discharge; up to 60 days.
  Mean number of days patients stayed in ICU
Length of hospitalization | From hospital admission to hospital discharge; up to 60 days.
  Mean number of days patients stayed at the hospital
Duration of invasive mechanical ventilation (IMV) | From first day patient are mechanically ventilated to IMV stop; up to 60 days.
  Mean number of days patients were invasively mechanically ventilated
Patients returned home | Up to 60 days.
  Number of patients that following hospital discharge returned home
Patients discharged to in-patient rehabilitation | Up to 60 days.
  Number of patients that were discharged from acute hospital to in-patient rehabilitation
Patients transferred to other hospitals | Up to 60 days.
  Number of patients that following hospital discharge were transferred to other hospitals
Exitus | From ICU admission until date of death from any cause, assessed up to 60 days.
  Number of patients that died from any cause during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Privitera, MSC, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Department of Pathophysiology and Transplantation, University of Milan Internal Medicine Department, Respiratory Unit and Cystic Fibrosis Adult Center, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Result] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Result] Kim RY, Murphy TE, Doyle M, Pulaski C, Singh M, Tsang S, Wicker D, Pisani MA, Connors GR, Ferrante LE. Factors Associated With Discharge Home Among Medical ICU Patients in an Early Mobilization Program. Crit Care Explor. 2019 Nov 11;1(11):e0060. doi: 10.1097/CCE.0000000000000060. eCollection 2019 Nov. PMID 32166241
- [Result] Lazzeri M, Lanza A, Bellini R, Bellofiore A, Cecchetto S, Colombo A, D'Abrosca F, Del Monaco C, Gaudiello G, Paneroni M, Privitera E, Retucci M, Rossi V, Santambrogio M, Sommariva M, Frigerio P. Respiratory physiotherapy in patients with COVID-19 infection in acute setting: a Position Paper of the Italian Association of Respiratory Physiotherapists (ARIR). Monaldi Arch Chest Dis. 2020 Mar 26;90(1). doi: 10.4081/monaldi.2020.1285. PMID 32236089